CLINICAL TRIAL: NCT00181779
Title: Open-Label Pilot Study of Aripiprazole for the Treatment of Mania in Children and Adolescents With Bipolar I, Bipolar II, and Bipolar Spectrum Disorder
Brief Title: Aripiprazole for the Treatment of Mania in Children and Adolescents With Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Joseph Biederman, MD, Chief, Clinical and Research Program in Pediatric Psychopharmacology and Adult ADHD; Professor of Psychiatry, Harvard Medical School, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-P-000153
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Bipolar Disorder; Mania
Keywords: mania; Abilify; children; bipolar disorder
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — Aripiprazole

INTERVENTIONS:
Drug: aripiprazole (Abilify)

SUMMARY:
This is an open-labeled study of Aripiprazole, testing its efficacy in the treatment of mania in children and adolescents with Bipolar I, Bipolar II and Bipolar Spectrum Disorder over 8 weeks. This is an exploratory, pilot study, seeking to determine whether Aripiprazole is efficacious and well tolerated in the treatment of youth with pediatric bipolar and bipolar spectrum disorder. The study results will be used to generate hypotheses for a larger randomized controlled clinical trial with explicit hypotheses and sufficient statistical power.

DETAILED DESCRIPTION:
Initial clinical evidence suggests that atypical neuroleptics may play a unique therapeutic role in the management of pediatric bipolar disorder. Aripiprazole is a novel neuroleptic recently approved by the FDA for the treatment of schizophrenia, and it has a unique pharmacological profile believed to be fundamentally different from other available antipsychotics. Many previous studies have reported increased efficacy of Aripiprazole compared to placebo. Unfortunately, Aripiprazole has not been investigated in children and adolescents, and as such, safety and efficacy has not been established for these populations.

This is an exploratory, pilot study, seeking to determine whether Aripiprazole is efficacious and well tolerated in the treatment of youth with pediatric bipolar and bipolar spectrum disorder. The study results, gathered from an 8 week open-label treatment period and subsequent 10 month extension period, will be used to generate hypotheses for a larger randomized controlled clinical trial with explicit hypotheses and sufficient statistical power.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, 6-17 years of age.
2. Patient and parent must have a level of understanding sufficient to communicate intelligently with the investigator and study coordinator, and to cooperate with all tests and examinations required by the protocol.
3. Patients and their legal representative must be considered reliable.
4. Each patient and his/her authorized legal representative must understand the nature of the study. The patient's authorized legal representative must sign an informed consent document and the patient must sign an informed assent document.
5. Patient must have a diagnosis of bipolar I or bipolar II disorder and currently display an acute manic, hypomanic, or mixed episode (with or without psychotic features) according to the DSM-IV based on clinical assessment and confirmed by structured diagnostic interview (Kidd Schedule of Affective Disorders). Eligible will also be children with bipolar spectrum disorder (or sub-threshold bipolar disorder) operationalized as having severe mood disturbance, which meets DSM-IV Criteria A for bipolar disorder but meet fewer elements in criteria B (only require 2 items for elation category and 3 for irritability).
6. Patients must have an initial score on the Y-MRS total score of at least 15.
7. Patient must be able to participate in mandatory blood draws.
8. Patient must be able to swallow pills.

Exclusion Criteria:

1. Investigator and his/her immediate family; defined as the investigator's spouse, parent, child, grandparent, or grandchild.
2. Serious, unstable illness including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.
3. Uncorrected hypothyroidism or hyperthyroidism.
4. History of severe allergies or multiple adverse drug reactions.
5. Non-febrile seizures without a clear and resolved etiology.
6. Leukopenia or history of leukopenia without a clear and resolved etiology.
7. DSM-IV substance (except nicotine or caffeine) dependence within past 6 months.
8. Judged clinically to be at serious suicidal risk.
9. Any other concomitant medication with primarily central nervous system activity other than specified in Concomitant Medication portion of the protocol.
10. History of intolerance or a non-responder to Aripiprazole as determined by the clinician.
11. Treatment with nonreversible monoamine oxidase inhibitors within 2 weeks prior to Visit 2.
12. Current diagnosis of schizophrenia.
13. For concomitant stimulant therapy used to treat ADHD, patients must have been on a stable dose of the medication for 1 month prior to randomization.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20
Dates: Start 2003-02; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Scores on the Young Mania Rating Scales

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Biederman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States

REFERENCES:
- [Derived] Biederman J, Mick E, Spencer T, Doyle R, Joshi G, Hammerness P, Kotarski M, Aleardi M, Wozniak J. An open-label trial of aripiprazole monotherapy in children and adolescents with bipolar disorder. CNS Spectr. 2007 Sep;12(9):683-9. doi: 10.1017/s1092852900021519. PMID 17805214